CLINICAL TRIAL: NCT05520762
Title: Hospital Airway Resuscitation Trial: A Cluster-Randomized, Pragmatic Trial
Brief Title: Hospital Airway Resuscitation Trial
Acronym: HART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021-13691; R33HL162980 (NIH)
Record Dates: First submitted 2022-08-22; First posted 2022-08-30 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Arrest; Respiratory Failure
Keywords: Cardiac Arrest; Emergency Airway Management; In-hospital Cardiac Arrest; Endotracheal Intubation; Supraglottic Airway
MeSH Terms: conditions — Heart Arrest; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Cluster-randomized design with crossover
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First choice supraglottic airway device, Then First choice endotracheal intubation (Experimental): A strategy of 'first choice' supraglottic airway during cardiac arrest. Clinicians can deviate to the airway management approach of their choice if deemed to be in the best interest of the patient. As part of a cluster-randomized design, hospitals (4 in the system) will be assigned to one arm for a month and then cross-over to the other arm.
  Interventions: Procedure: A strategy of first choice supraglottic airway; Procedure: A strategy of first choice endotracheal intubation
- First choice endotracheal intubation, Then First choice supraglottic airway (Active Comparator): A strategy of 'first choice' endotracheal intubation during cardiac arrest. Clinicians can deviate to the airway management approach of their choice if deemed to be in the best interest of the patient. As part of a cluster-randomized design, hospitals (4 in the system) will be assigned to one arm for a month and then cross-over to the other arm.
  Interventions: Procedure: A strategy of first choice supraglottic airway; Procedure: A strategy of first choice endotracheal intubation

INTERVENTIONS:
Procedure: A strategy of first choice supraglottic airway — See description in Arms section
Procedure: A strategy of first choice endotracheal intubation — See description in Arms section

SUMMARY:
The Hospital Airway Resuscitation Trial (HART) is a cluster-randomized, pragmatic trial of advanced airway management with a strategy of first choice supraglottic airway vs. first choice endotracheal intubation during in-hospital cardiac arrest.

DETAILED DESCRIPTION:
In-hospital cardiac arrest occurs in nearly 300,000 hospitalized patients in the United States each year and results in substantial morbidity and mortality. Nevertheless, the evidence base guiding the management of in-hospital cardiac arrest is quite limited and society guidelines generally extrapolate data from the out-of-hospital cardiac setting to inform in-hospital arrest care. As compared to out-of-hospital arrest, however, in-hospital arrest victims tend to have more medical comorbidities, have a witnessed arrest, and be attended to by professional first responders with advanced monitoring and treatment capabilities. Advanced airway management is a key element of cardiac arrest resuscitation. The American Heart Association makes broad recommendations regarding airway management during in-hospital cardiac, supporting endotracheal intubation (a complex procedure requiring placement of an endotracheal tube through the vocal cords) and supraglottic airway placement (a less complex advanced airway modality wherein the device is placed blindly in the supraglottic space). Data from the out-of-hospital cardiac arrest setting has found that a supraglottic airway strategy may be similar or superior to a more complex endotracheal intubation strategy. There is no randomized data to guide practice in the in-hospital setting. We intend to address this knowledge gap by performing the Hospital Airway Resuscitation Trial (HART)-a highly-innovative, pragmatic cluster-randomized trial leveraging the unified clinical and research infrastructure within the Montefiore HealthSystem (New York City) to conduct a first-of-its-kind in-hospital arrest trial in a highly diverse patient population. Specifically, a mixture of academic and community hospitals within the MontefioreHealth system will be randomized to either a strategy of first-choice endotracheal intubation or a strategy of first choice supraglottic airway, with crossovers occurring at regular intervals. Key outcomes for the trial will include return of spontaneous circulation, alive-and-ventilator-free days, and hospital survival.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged >=18 years
2. Admitted to the hospital for any condition
3. Suffered in-hospital cardiac arrest (loss of pulse and ≥2 minutes of chest compressions)
4. Need for assisted ventilation (defined by initiation of bag-mask-ventilation or other supported ventilation)

Exclusion Criteria:

1. Cardiac arrest in the Operating Room or other area not responded to by Critical Care/Emergency Department (ED) teams.
2. Cardiac arrest in which an invasive airway (i.e. endotracheal tube, tracheostomy tube) is already in place
3. Patients with Do Not Resuscitate or Do Not Intubate orders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Alive-and-ventilator free days | From cardiac arrest until 28-days after cardiac arrest
  The number of days a patient is alive and breathing independently of invasive mechanical ventilation will be summarized by study arm using basic descriptive statistics. A patient who leaves the hospital alive and is not discharged to a hospice setting, will be considered to have lived to 28-days. A patient discharged to a hospice facility will be assessed as having died on the day of hospital discharge. A patient who is discharged on invasive mechanical ventilation, will be assumed to have remained on invasive mechanical ventilation through 28-days.

SECONDARY OUTCOMES:
Return of spontaneous circulation (ROSC) | Onset of in-hospital cardiac arrest event until either ROSC or death up to 24 hours
  ROSC will be assessed. ROSC is defined as having ≥20 minutes of continuous spontaneous circulation without chest compressions. Rates of ROSC will be summarized by study arm using basic descriptive statistics.
72 hour survival | From IHCA event until 72 hours after IHCA event
  Survival to 72 hour after in-hospital cardiac arrest (IHCA) event will be summarized by study arm using basic descriptive statistics.
28 day survival | From IHCA event until 28 days after IHCA event
  Survival to 28 days after cardiac IHCA event will be summarized by study arm using basic descriptive statistics.
Functional Outcome at Discharge | Time of hospital discharge
  Functional Outcome at Discharge will be measured using the modified Rankin Scale (mRS). The mRS is a clinical tool that measures the patient's function disability (ability to perform daily living activities). The mRS is based on a 7-point scale ranging from 0 ("No symptoms at all") to 6 ("Death") such that higher scores are associated with increased functional disability. Scores at discharge can be used as a proxy to help identify patients who may require closer follow-up given the difficulty in obtaining long-term follow-up. mRS scores will be dichotomized to identify all patients with mRS>3 and summarized by study arm.
Survival to hospital discharge | From IHCA event until 60 days after cardiac arrest
  Survival to hospital discharge, truncated at 60 days for the purposes of this outcome, will be summarized by study arm using basic descriptive statistics.

OTHER OUTCOMES:
Prolonged pauses | From start of chest compressions during cardiac arrest until ROSC or death up to 24-hours
  The number of prolonged pauses, defined as pauses lasting >5 seconds in duration, in chest compressions during active Cardiopulmonary Resuscitation (CPR) will be determined. Prolonged pauses will be summarized by study arm using basic descriptive statistics.
Rate of ventilator-associated pneumonia (VAP) | Cardiac arrest until 7 days after cardiac arrest
  Rate of VAP in the 7 days after cardiac arrest. VAP defined as new pneumonia while receiving mechanical ventilation after cardiac arrest. New pneumonia will be defined by 1) new pulmonary infiltrate on chest imaging 2) either new/worsening fever or leukocytosis 3) either change in sputum composition/frequency or worsening gas exchange or new/worsening cough or dyspnea. Rates of VAP will be summarized by study arm using basic descriptive statistics.
Chest compression fraction | From start of chest compressions during cardiac arrest until ROSC or death up to 24-hours
  Percentage of total cardiac arrest time during which chest compressions are being performed will be determined. Results will be summarized by study arm using basic descriptive statistics.
Time to advanced airway | Time from initiation of chest compressions to advanced airway placement
  Time from initiation of chest compressions to advanced airway placement
Longest Overall Pause in Chest Compression | At time of cardiac arrest, less than one day
  The duration of the longest overall pause in chest compression will be determined. This interval will be summarized by arm using basic descriptive statistics. It is hypothesized that supraglottic airway (SGA) placement will result in chest compression pauses of shorter durations.
Number of Overall Pauses in Chest Compression | At time of cardiac arrest, less than one day
  The number of overall pauses in chest compression, greater than 5 seconds in duration, will be summarized by arm using basic descriptive statistics. It is hypothesized that SGA placement will result in fewer chest compression pauses
Time to epinephrine | Time from initiation of chest compressions to first epinephrine for cardiac arrest with initial non-shockable rhythm
  Time from initiation of chest compressions to first epinephrine for cardiac arrest with initial non-shockable rhythm

CONTACTS AND LOCATIONS:
Overall Officials: Ari Moskowitz, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Holmberg MJ, Ross CE, Fitzmaurice GM, Chan PS, Duval-Arnould J, Grossestreuer AV, Yankama T, Donnino MW, Andersen LW; American Heart Association's Get With The Guidelines-Resuscitation Investigators. Annual Incidence of Adult and Pediatric In-Hospital Cardiac Arrest in the United States. Circ Cardiovasc Qual Outcomes. 2019 Jul 9;12(7):e005580. PMID 31545574
- [Background] Coute RA, Panchal AR, Mader TJ, Neumar RW. National Institutes of Health-Funded Cardiac Arrest Research: A 10-Year Trend Analysis. J Am Heart Assoc. 2017 Jul 12;6(7):e005239. doi: 10.1161/JAHA.116.005239. PMID 28701308
- [Background] Sinha SS, Sukul D, Lazarus JJ, Polavarapu V, Chan PS, Neumar RW, Nallamothu BK. Identifying Important Gaps in Randomized Controlled Trials of Adult Cardiac Arrest Treatments: A Systematic Review of the Published Literature. Circ Cardiovasc Qual Outcomes. 2016 Nov;9(6):749-756. doi: 10.1161/CIRCOUTCOMES.116.002916. Epub 2016 Oct 18. PMID 27756794
- [Background] Wang HE, Kupas DF, Greenwood MJ, Pinchalk ME, Mullins T, Gluckman W, Sweeney TA, Hostler D. An algorithmic approach to prehospital airway management. Prehosp Emerg Care. 2005 Apr-Jun;9(2):145-55. doi: 10.1080/10903120590924618. PMID 16036838
- [Background] Panchal AR, Bartos JA, Cabanas JG, Donnino MW, Drennan IR, Hirsch KG, Kudenchuk PJ, Kurz MC, Lavonas EJ, Morley PT, O'Neil BJ, Peberdy MA, Rittenberger JC, Rodriguez AJ, Sawyer KN, Berg KM; Adult Basic and Advanced Life Support Writing Group. Part 3: Adult Basic and Advanced Life Support: 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2020 Oct 20;142(16_suppl_2):S366-S468. doi: 10.1161/CIR.0000000000000916. Epub 2020 Oct 21. No abstract available. PMID 33081529
- [Background] Bradley SM, Zhou Y, Ramachandran SK, Engoren M, Donnino M, Girotra S. Retrospective cohort study of hospital variation in airway management during in-hospital cardiac arrest and the association with patient survival: insights from Get With The Guidelines-Resuscitation. Crit Care. 2019 May 6;23(1):158. doi: 10.1186/s13054-019-2426-5. PMID 31060580
- [Background] Wang HE, Schmicker RH, Daya MR, Stephens SW, Idris AH, Carlson JN, Colella MR, Herren H, Hansen M, Richmond NJ, Puyana JCJ, Aufderheide TP, Gray RE, Gray PC, Verkest M, Owens PC, Brienza AM, Sternig KJ, May SJ, Sopko GR, Weisfeldt ML, Nichol G. Effect of a Strategy of Initial Laryngeal Tube Insertion vs Endotracheal Intubation on 72-Hour Survival in Adults With Out-of-Hospital Cardiac Arrest: A Randomized Clinical Trial. JAMA. 2018 Aug 28;320(8):769-778. doi: 10.1001/jama.2018.7044. PMID 30167699
- [Background] Moskowitz A, Holmberg MJ, Donnino MW, Berg KM. In-hospital cardiac arrest: are we overlooking a key distinction? Curr Opin Crit Care. 2018 Jun;24(3):151-157. doi: 10.1097/MCC.0000000000000505. PMID 29688939
- [Background] Apfelbaum JL, Hagberg CA, Connis RT, Abdelmalak BB, Agarkar M, Dutton RP, Fiadjoe JE, Greif R, Klock PA, Mercier D, Myatra SN, O'Sullivan EP, Rosenblatt WH, Sorbello M, Tung A. 2022 American Society of Anesthesiologists Practice Guidelines for Management of the Difficult Airway. Anesthesiology. 2022 Jan 1;136(1):31-81. doi: 10.1097/ALN.0000000000004002. PMID 34762729
- [Background] Yehya N, Harhay MO, Curley MAQ, Schoenfeld DA, Reeder RW. Reappraisal of Ventilator-Free Days in Critical Care Research. Am J Respir Crit Care Med. 2019 Oct 1;200(7):828-836. doi: 10.1164/rccm.201810-2050CP. PMID 31034248
- [Background] Schoenfeld DA, Bernard GR; ARDS Network. Statistical evaluation of ventilator-free days as an efficacy measure in clinical trials of treatments for acute respiratory distress syndrome. Crit Care Med. 2002 Aug;30(8):1772-7. doi: 10.1097/00003246-200208000-00016. PMID 12163791
- [Background] Witten L, Gardner R, Holmberg MJ, Wiberg S, Moskowitz A, Mehta S, Grossestreuer AV, Yankama T, Donnino MW, Berg KM. Reasons for death in patients successfully resuscitated from out-of-hospital and in-hospital cardiac arrest. Resuscitation. 2019 Mar;136:93-99. doi: 10.1016/j.resuscitation.2019.01.031. Epub 2019 Jan 30. PMID 30710595
- [Background] Haywood K, Whitehead L, Nadkarni VM, Achana F, Beesems S, Bottiger BW, Brooks A, Castren M, Ong MEH, Hazinski MF, Koster RW, Lilja G, Long J, Monsieurs KG, Morley PT, Morrison L, Nichol G, Oriolo V, Saposnik G, Smyth M, Spearpoint K, Williams B, Perkins GD; COSCA Collaborators. COSCA (Core Outcome Set for Cardiac Arrest) in Adults: An Advisory Statement From the International Liaison Committee on Resuscitation. Resuscitation. 2018 Jun;127:147-163. doi: 10.1016/j.resuscitation.2018.03.022. Epub 2018 Apr 26. PMID 29706235
- [Background] Hemming K, Kasza J, Hooper R, Forbes A, Taljaard M. A tutorial on sample size calculation for multiple-period cluster randomized parallel, cross-over and stepped-wedge trials using the Shiny CRT Calculator. Int J Epidemiol. 2020 Jun 1;49(3):979-995. doi: 10.1093/ije/dyz237. PMID 32087011
- [Background] Sevransky JE, Rothman RE, Hager DN, Bernard GR, Brown SM, Buchman TG, Busse LW, Coopersmith CM, DeWilde C, Ely EW, Eyzaguirre LM, Fowler AA, Gaieski DF, Gong MN, Hall A, Hinson JS, Hooper MH, Kelen GD, Khan A, Levine MA, Lewis RJ, Lindsell CJ, Marlin JS, McGlothlin A, Moore BL, Nugent KL, Nwosu S, Polito CC, Rice TW, Ricketts EP, Rudolph CC, Sanfilippo F, Viele K, Martin GS, Wright DW; VICTAS Investigators. Effect of Vitamin C, Thiamine, and Hydrocortisone on Ventilator- and Vasopressor-Free Days in Patients With Sepsis: The VICTAS Randomized Clinical Trial. JAMA. 2021 Feb 23;325(8):742-750. doi: 10.1001/jama.2020.24505. PMID 33620405
- [Background] Nichol G, Brown SP, Perkins GD, Kim F, Sterz F, Broeckel Elrod JA, Mentzelopoulos S, Lyon R, Arabi Y, Castren M, Larsen P, Valenzuela T, Graesner JT, Youngquist S, Khunkhlai N, Wang HE, Ondrej F, Sastrias JM, Barasa A, Sayre MR. What change in outcomes after cardiac arrest is necessary to change practice? Results of an international survey. Resuscitation. 2016 Oct;107:115-20. doi: 10.1016/j.resuscitation.2016.08.004. Epub 2016 Aug 23. PMID 27565860
- [Background] Moskowitz A, Andrea L, Shiloh AL, Cardasis J, Carty C, Kim M, Xie X, McAllen S, Esses D, Lutz C, Takematsu M, Romero J, Schimmrich K, Fein DG, Dodi AE, Rednor S, Bangar M, Mohamed A, Eisen LA, Wang HE, Donnino MW, Gong MN. Design and implementation of the hospital airway resuscitation trial. Resusc Plus. 2023 Nov 30;17:100512. doi: 10.1016/j.resplu.2023.100512. eCollection 2024 Mar. PMID 38076388
- [Background] Fein DG, Zhao D, Swartz K, Nauka P, Andrea L, Aboodi M, Shiloh AL, Eisen LA. The Impact of Nighttime on First Pass Success During the Emergent Endotracheal Intubation of Critically Ill Patients. J Intensive Care Med. 2021 Dec;36(12):1498-1506. doi: 10.1177/0885066620965166. Epub 2020 Oct 15. PMID 33054483
- [Background] Nauka PC, Chen JT, Shiloh AL, Eisen LA, Fein DG. Practice, Outcomes, and Complications of Emergent Endotracheal Intubation by Critical Care Practitioners During the COVID-19 Pandemic. Chest. 2021 Dec;160(6):2112-2122. doi: 10.1016/j.chest.2021.06.008. Epub 2021 Jun 15. PMID 34139207
- [Background] Janz DR, Semler MW, Lentz RJ, Matthews DT, Assad TR, Norman BC, Keriwala RD, Ferrell BA, Noto MJ, Shaver CM, Richmond BW, Zinggeler Berg J, Rice TW; Facilitating EndotracheaL intubation by Laryngoscopy technique and apneic Oxygenation Within the ICU Investigators and the Pragmatic Critical Care Research Group. Randomized Trial of Video Laryngoscopy for Endotracheal Intubation of Critically Ill Adults. Crit Care Med. 2016 Nov;44(11):1980-1987. doi: 10.1097/CCM.0000000000001841. PMID 27355526
- [Background] Driver B, Dodd K, Klein LR, Buckley R, Robinson A, McGill JW, Reardon RF, Prekker ME. The Bougie and First-Pass Success in the Emergency Department. Ann Emerg Med. 2017 Oct;70(4):473-478.e1. doi: 10.1016/j.annemergmed.2017.04.033. PMID 28601269
- [Background] Driver BE, Prekker ME, Klein LR, Reardon RF, Miner JR, Fagerstrom ET, Cleghorn MR, McGill JW, Cole JB. Effect of Use of a Bougie vs Endotracheal Tube and Stylet on First-Attempt Intubation Success Among Patients With Difficult Airways Undergoing Emergency Intubation: A Randomized Clinical Trial. JAMA. 2018 Jun 5;319(21):2179-2189. doi: 10.1001/jama.2018.6496. PMID 29800096
- [Background] Driver BE, Semler MW, Self WH, Ginde AA, Trent SA, Gandotra S, Smith LM, Page DB, Vonderhaar DJ, West JR, Joffe AM, Mitchell SH, Doerschug KC, Hughes CG, High K, Landsperger JS, Jackson KE, Howell MP, Robison SW, Gaillard JP, Whitson MR, Barnes CM, Latimer AJ, Koppurapu VS, Alvis BD, Russell DW, Gibbs KW, Wang L, Lindsell CJ, Janz DR, Rice TW, Prekker ME, Casey JD; BOUGIE Investigators and the Pragmatic Critical Care Research Group. Effect of Use of a Bougie vs Endotracheal Tube With Stylet on Successful Intubation on the First Attempt Among Critically Ill Patients Undergoing Tracheal Intubation: A Randomized Clinical Trial. JAMA. 2021 Dec 28;326(24):2488-2497. doi: 10.1001/jama.2021.22002. PMID 34879143
- [Background] Self WH, Semler MW, Wanderer JP, Ehrenfeld JM, Byrne DW, Wang L, Atchison L, Felbinger M, Jones ID, Russ S, Shaw AD, Bernard GR, Rice TW. Saline versus balanced crystalloids for intravenous fluid therapy in the emergency department: study protocol for a cluster-randomized, multiple-crossover trial. Trials. 2017 Apr 13;18(1):178. doi: 10.1186/s13063-017-1923-6. PMID 28407811
- [Background] Semler MW, Self WH, Wanderer JP, Ehrenfeld JM, Wang L, Byrne DW, Stollings JL, Kumar AB, Hughes CG, Hernandez A, Guillamondegui OD, May AK, Weavind L, Casey JD, Siew ED, Shaw AD, Bernard GR, Rice TW; SMART Investigators and the Pragmatic Critical Care Research Group. Balanced Crystalloids versus Saline in Critically Ill Adults. N Engl J Med. 2018 Mar 1;378(9):829-839. doi: 10.1056/NEJMoa1711584. Epub 2018 Feb 27. PMID 29485925
- [Background] Gong MN, Schenk L, Gajic O, Mirhaji P, Sloan J, Dong Y, Festic E, Herasevich V. Early intervention of patients at risk for acute respiratory failure and prolonged mechanical ventilation with a checklist aimed at the prevention of organ failure: protocol for a pragmatic stepped-wedged cluster trial of PROOFCheck. BMJ Open. 2016 Jun 10;6(6):e011347. doi: 10.1136/bmjopen-2016-011347. PMID 27288382
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- See also: International Committee of Medical Journal Editors. Defining the Role of Authors and Contributors. Accessed July 6, 2017. — http://www.icmje.org/recommendations/browse/roles-and-responsibilities/defining-the-role-of-authors-and-contributors.html